CLINICAL TRIAL: NCT06609967
Title: Effect of Autologous Platelet Rich Fibrin (PRF) on Post-Operative Complications and Healing Following the Extractions Impacted Mandibular Wisdoms
Brief Title: Effect of Autologous Platelet Rich Fibrin on Post-Operative Complications and Healing Following the Extraction
Acronym: PRF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dow University of Health Sciences (Other)
Responsible Party: Principal Investigator, Hamza Jawed, Principal Investigator, Dow University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Hamza001
Record Dates: First submitted 2021-08-27; First posted 2024-09-24 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-09

CONDITIONS: Pain, Postoperative; Post Operative Swelling; Trismus; Soft Tissue Healing
Keywords: prf; extraction socket; post operative complications; wisdom tooth extractions; surgical extractions
MeSH Terms: conditions — Pain, Postoperative; Trismus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PRF group (Experimental)
  Interventions: Procedure: application of PRF
- Non-PRF group (Active Comparator)
  Interventions: Procedure: application of conventional surgicel

INTERVENTIONS:
Procedure: application of PRF — PRF will be randomly administered into one group of patients undergoing any extractions group A (Right after the extraction) Group B will be a control group in which extraction sockets will be left to heal with the natural blood clot. Consenting patients will be assigned into groups randomly and not informed which group they were placed into. The PRF will be administered obtained from a tube of 10 ml blood and no material will be placed in the control group. The progress of healing and post-operative complications will be tracked over a period of 7 days with patients being called for follow-up on days 3, 5 and 7
  Arms: PRF group
Procedure: application of conventional surgicel — it will be a control group in which extraction sockets will be left to heal with the natural blood clot.
  Arms: Non-PRF group

SUMMARY:
As post-operative pain, infection inflammation and infections are the main complications after the surgical extraction of the lower third molar the aim of this study is to compare the healing effects of PRF administered postoperatively

DETAILED DESCRIPTION:
PRF will be randomly administered into one group of patients undergoing any extractions group A (Right after the extraction) Group B will be a control group in which extraction sockets will be left to heal with the natural blood clot. Consenting patients will be assigned into groups randomly and not informed which group they were placed into. The PRF will be administered obtained from a tube of 10 ml blood and no material will be placed in the control group. The progress of healing and post-operative complications will be tracked over a period of 7 days with patients being called for follow-up on days 3, 5 and 7. Their post-operative complications will be checked at every subsequent visit and noted in the questionnaire. The Questionnaire is structured and will be interviewer-administered. It will comprise of basic bio-demographic data (such as name, age, sex, etc) and 3 closed-ended questions related to post-operative complications following the extraction

ELIGIBILITY:
Inclusion Criteria:

1. Both male and female patients
2. Patients that give their consent to the use of their information and to the administration of the drug will be the participants of the study.
3. Patients with 3rd molar impactions
4. Absence of systemic diseases
5. age ⩾18 years and the ability to cooperate with the requirements of the study protocol.

Exclusion Criteria:

1. Medically compromised patients.
2. Immunocompromised patients.
3. Patients that do not consent.
4. Patients that are below the age of 17.
5. Patients that are pregnant.
6. Fully erupted molars will be excluded. smokers (> 5 a day) will be excluded as well.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
Pain | 7 days
  Post-operative pain will be measured using a visual analog scale in both groups i.e. conventional therapy group and PRF group on the 1st, 3rd and 7th post operative day.
Post operative Swelling | 7 days
  Post operative swelling will be measured in terms of metric calculation (centimeters) in 2 sites i.e: 1. From the tragus of the ear to angle of mouth and 2. From lateral canthus of eye to angle of mandible on the 3rd and 7th post operative day.
Trismus- Post surgical limitation in mouth opening | 7 days
  Trismus will be measured as the distance in (cm) between the edges of the maxillary and mandibular central incisors post surgically on the 3rd and 7th post operative day.
Wound/ extraction socket healing | 7 days
  The wound healing of the extraction socket of mandibular wisdom teeth will be assessed according to Landry's criteria on the 7th post operative day.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Oral and Maxillofacial Surgery, Dow University of Health Sciences, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided
Complete data will be shared after consent.

REFERENCES:
- [Background] Passarelli PC, Romeo A, Lopez MA, De Angelis P, Desantis V, Piccirillo GB, Papa R, Papi P, Pompa G, Moffa A, Casale M, D'Addona A. Evaluation of the periodontal healing of the second mandibular molar distal site following insertion of PRF in the third molar post extraction alveolus. J Biol Regul Homeost Agents. 2020 Sep-Oct;34(5 Suppl. 3):111-118. Technology in Medicine. PMID 33386040